CLINICAL TRIAL: NCT03364959
Title: Ex Vivo Pilot Study of the Impact of Nasal Breathing During the Administration of Inhaled Corticosteroids by Inhalation Chamber in Asthmatic Children Ages Between 1 and 4-year-old
Acronym: MASQUE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016-47; 2016-A01839-42 (Other: ANSM)
Record Dates: First submitted 2017-11-06; First posted 2017-12-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flixotide (Experimental): Patients inhale first Flixotide and then Qvar
  Interventions: Other: Corticosteroids inhalation
- Qvar (Experimental): Patients inhale first Qvar and then Flixotide
  Interventions: Other: Corticosteroids inhalation

INTERVENTIONS:
Other: Corticosteroids inhalation — Flixotide inhalation followed by Qvar inhalation through a nasal filter and a mouth filter located in a partitioned face mask and delivered to an infant with asthma via a Tipshaler® holding chamber
  Arms: Flixotide
Other: Corticosteroids inhalation — Qvar inhalation followed by Flixotide inhalation through a nasal filter and a mouth filter located in a partitioned face mask and delivered to an infant with asthma via a Tipshaler® holding chamber
  Arms: Qvar

SUMMARY:
The main purpose of this open randomized, ex-vivo comparative study, is to assess and to compare the inhalable dose of inhaled corticosteroid collected through a nasal filter and a mouth filter located in a partitioned face mask and delivered to an infant with asthma via a Tipshaler® holding chamber

DETAILED DESCRIPTION:
The use of a face mask is recommended for inhaled treatments delivered from a pressurized metered-dose inhaler and a spacer device in infants and young children with respiratory disorders such as asthma.

The nose effectively filters the air particles and it may reduce the amount of inhaled drug. Thus it is reported that the drug deposited in the lung dose is halved in older children inhaling through the nose with respect to those inhaling through the mouth.

In very young children the efficiency of nasal filtration is unknown for inhaled treatment. In infants, an in-vitro study suggests that nasal breathing allows a similar or more important drug delivery than mouth breathing, contrary to what is observed in the oldest and adults.

So it seems of great import to characterize the drug delivery in this age group comparing the nasal with the mouth breathing.

The main purpose of this open randomized, ex-vivo comparative study, is to assess and to compare the inhalable dose of inhaled corticosteroid collected through a nasal filter and a mouth filter located in a partitioned face mask and delivered to an infant with asthma via a Tipshaler® holding chamber. 60 children, aged between 1 and 4 years old, with a medically diagnosed asthma will be recruited. Each child will inhale four puffs of both Fluticasone 125 µg/puff and Beclometasone dipropionate 100 µg/puff administered by a single observer in a standardized and randomized way. No drug will be inhaled by the children. The drugs collected on the filters between the holding chamber and patient will be analysed by high performance liquid chromatography HPLC). Filter doses will be expressed in percentage of the total dose filtered. The analysis will cover the difference between oral dose and nasal dose compared to zero. Student's test will be performed with p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 1 to 4 years old
* Male or female
* With medically diagnosed asthma
* Patients who are used to use an inhalation chamber with a face mask
* Patients who have not had asthmatic decompensation for at least 1 month.
* Patients' parents having given their written consent
* With normal clinical respiratory examination on the day of the test.

Exclusion Criteria:

* Patients whose parents are unable to understand the purpose and conditions of the study
* Patients whose parents are unable to give their consent
* Patients participating in another clinical trial or exclusion period from a previous clinical trial
* Patients presenting with a nasopharyngeal infection in the previous month
* Child with nasal obstruction, nocturnal snoring, adenoid facies or facial malformation
* Patient presenting with an asthmatic decompensation episode in the previous month

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of corticoisteroids proportion delivered to the nose with respect to the mouth by chromatography. | 12 months
  Compare by chromatography the proportion of product administered to the nose with respect to the mouth for the administration of inhaled corticosteroids in children with asthma. Filter doses will be expressed as a percentage of the total filtered dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided